CLINICAL TRIAL: NCT02694328
Title: A Phase 3 Study to Evaluate Weight Gain of ALKS 3831 Compared to Olanzapine in Adults With Schizophrenia
Brief Title: A Study of ALKS 3831 in Adults With Schizophrenia (The ENLIGHTEN-2 Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK3831-A303
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia
Keywords: Alkermes; ALKS 3831; Samidorphan; Schizophrenia; Olanzapine; Weight
MeSH Terms: conditions — Schizophrenia; Body Weight | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALKS 3831 (Experimental): Administered as a coated bilayer tablet
  Interventions: Drug: ALKS 3831
- Olanzapine (Active Comparator): Administered as a coated bilayer tablet
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: ALKS 3831 — Daily dosing
  Arms: ALKS 3831
Drug: Olanzapine — Daily dosing
  Arms: Olanzapine

SUMMARY:
This study will evaluate weight gain of ALKS 3831 compared to olanzapine in adult subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) of 18.0-30.0 kg/m^2, inclusive, at Visit 1 and Visit 2
* Subject meets the DSM-5 criteria for a primary diagnosis of schizophrenia
* Subject is appropriate for outpatient treatment; has no hospitalizations for acute exacerbations of schizophrenia within 6 months before Visit 1
* Subject has maintained a stable body weight (change </= 5%) for at least 3 months prior to Visit 1 based on self-report
* Additional criteria may apply

Exclusion Criteria:

* Subject has any of the following psychiatric conditions per DSM-5 criteria:
* Diagnosis of schizoaffective disorder or bipolar I or II disorder, or current, untreated or unstable major depressive disorder
* Clinically significant cognitive difficulties present within the past 2 years that could interfere with participation in the study
* Drug-induced or toxic psychosis
* Any other psychiatric condition that could interfere with participation in the study
* Subject poses a current suicide risk at Visit 1 or Visit 2 in the opinion of the investigator
* Subject has inflammatory bowel disease or any other gastrointestinal disorder associated with weight loss, anorexia nervosa, or binge eating disorder
* Additional criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 561 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Study Director — Alkermes, Inc.
Locations (50):
- United States (49):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Springdale, Arkansas
  - Alkermes Investigational Site, Anaheim, California
  - Alkermes Investigational Site, Cerritos, California
  - Alkermes Investigational Site, Culver City, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Glendale, California
  - Alkermes Investigational Site, Long Beach, California
  - Alkermes Investigational Site, National City, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, Pico Rivera, California
  - Alkermes Investigational Site, Redlands, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Temecula, California
  - Alkermes Investigational Site, Torrance, California
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Lauderhill, Florida
  - Alkermes Investigational Site, Miami, Florida
  - Alkermes Investigational Site, North Miami, Florida
  - Alkermes Investigational Site, Oakland Park, Florida
  - Alkermes Investigational Site, Tampa, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Augusta, Georgia
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Grand Rapids, Michigan
  - Alkermes Investigational Site, Flowood, Mississippi
  - Alkermes Investigational Site, Creve Coeur, Missouri
  - Alkermes Investigational Site, O'Fallon, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Las Vegas, Nevada
  - Alkermes Investigational Site, Berlin, New Jersey
  - Alkermes Investigational Site, Marlton, New Jersey
  - Alkermes Investigational Site, Brooklyn, New York
  - Alkermes Investigational Site, Jamaica, New York
  - Alkermes Investigational Site, New York, New York
  - Alkermes Investigational Site, Rochester, New York
  - Alkermes Investigational Site, Wards Island, New York
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Middleburg Heights, Ohio
  - Alkermes Investigational Site, Allentown, Pennsylvania
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Bellevue, Washington
- Alkermes Investigational Site, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Correll CU, Stein E, Graham C, DiPetrillo L, Akerman S, Stanford AD, Jiang Y, Yagoda S, McDonnell D, Hopkinson C. Reduction in Multiple Cardiometabolic Risk Factors With Combined Olanzapine/Samidorphan Compared With Olanzapine: Post Hoc Analyses From a 24-Week Phase 3 Study. Schizophr Bull. 2023 Mar 15;49(2):454-463. doi: 10.1093/schbul/sbac144. PMID 36305696
- [Derived] Meyer JM, Simmons A, Jiang Y, Graham C, Yagoda S, McDonnell D. Olanzapine/samidorphan combination consistently mitigates weight gain across various subgroups of patients. CNS Spectr. 2023 Aug;28(4):478-481. doi: 10.1017/S1092852922000967. Epub 2022 Oct 13. PMID 36226902

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olanzapine | ALKS 3831
Started | 276 | 274
Completed | 176 | 176
Not Completed | 100 | 98
Not completed — Adverse Event | 27 | 33
Not completed — Withdrawal by Subject | 27 | 23
Not completed — Lost to Follow-up | 26 | 22
Not completed — Noncompliant with study drug | 11 | 8
Not completed — Incarceration | 1 | 1
Not completed — Lack of Efficacy | 1 | 2
Not completed — Pregnancy | 1 | 1
Not completed — Protocol Violation | 6 | 5
Not completed — Abnormal Laboratory Value | 0 | 3

BASELINE CHARACTERISTICS:
Population: Disposition is shown for the safety population - subjects who were randomized and received at least 1 dose of study drug. 5 subject in the olanzapine group and 6 subject in the ALKS 3831 group were randomized but not treated, and thus were not included in the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | ALKS 3831 | Total
Number analyzed (Participants) | 276 | 274 | 550
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.01) | 40.3 (9.79) | 40.2 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 81 | 150
  Male | 207 | 193 | 400
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 37 | 79
  Not Hispanic or Latino | 234 | 237 | 471
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 193 | 199 | 392
  White | 65 | 63 | 128
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 276 | 274 | 550

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight at Week 24
Time Frame: Baseline and Week 24
Population: The full analysis set (FAS) population includes all randomized subjects who received at least 1 dose of study drug and had at least 1 postbaseline weight assessment
Measure: Least Squares Mean (Standard Error); unit: Percent change in body weight
Arm/Group | Olanzapine | ALKS 3831
Number analyzed (Participants) | 272 | 266
Percent change in body weight | 6.59 (0.668) | 4.21 (0.681)
Statistical Analysis 1: Comparison: ALKS 3831; Test type: Superiority; p = 0.003, ANCOVA — P-value was adjusted using the Cui, Hung, and Wang (CHW) method to account for the unblinded interim analysis for sample size re-estimation; Missing values at Week 24 were imputed using multiple imputation; Least Squares Mean Difference = -2.38, 95% CI 2-sided [-3.88 to -0.88], Standard Error of Mean 0.765

2. Primary Outcome: Percentage of Participants With >/= 10% Weight Gain at Week 24
Time Frame: Baseline and Week 24
Population: The FAS population included all randomized subjects who received at least 1 dose of study drug and had at least 1 postbaseline weight assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Olanzapine | ALKS 3831
Number analyzed (Participants) | 272 | 266
Percentage of participants | 29.8 | 17.8
Statistical Analysis 1: Comparison: Olanzapine vs ALKS 3831; Test type: Superiority; p = 0.003, Regression, Logistic — P-value was adjusted using the CHW method to account for the unblinded interim analysis for sample size re-estimation; Missing values at Week 24 were imputed using multiple imputation; Risk Difference (RD) = -13.7, 95% CI 2-sided [-22.8 to -4.6] — Risk difference (RD) of ALKS 3831 vs. Olanzapine

3. Secondary Outcome: Percentage of Participants With >/= 7% Weight Gain at Week 24
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Olanzapine | ALKS 3831
Number analyzed (Participants) | 272 | 266
Percentage of participants | 42.7 | 27.5
Statistical Analysis 1: Comparison: Olanzapine vs ALKS 3831; Test type: Superiority; p = 0.001, Regression, Logistic; Missing values at Week 24 were imputed using multiple imputation; Risk Difference (RD) = -15.9, 95% CI 2-sided [-25.3 to -6.5] — Risk difference (RD) ALKS 3831 vs. Olanzapine

4. Secondary Outcome: Number of Participants Experiencing of Adverse Events (AEs)
Time Frame: 24 weeks
Population: The Safety Population includes all randomized subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine | ALKS 3831
Number analyzed (Participants) | 276 | 274
Participants | 227 | 203

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Arm/Group | Olanzapine | ALKS 3831
All-Cause Mortality (participants affected / at risk) | 0/276 | 0/274
Serious Adverse Events (participants affected / at risk) | 7/276 | 10/274
Other Adverse Events (participants affected / at risk) | 159/276 | 146/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=276) | ALKS 3831 (N=274)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 3 (3) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=276) | ALKS 3831 (N=274)
Dry mouth (Gastrointestinal disorders) | 22 (22) | 35 (36)
Extra dose administered (Injury, poisoning and procedural complications) | 17 (29) | 14 (18)
Weight increased (Investigations) | 100 (102) | 68 (68)
Waist circumference increased (Investigations) | 22 (22) | 17 (17)
Blood creatine phosphokinase increased (Investigations) | 12 (15) | 14 (16)
Increased appetite (Metabolism and nutrition disorders) | 34 (35) | 30 (30)
Somnolence (Nervous system disorders) | 50 (57) | 58 (63)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02694328/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02694328/SAP_001.pdf